CLINICAL TRIAL: NCT04108728
Title: Neuropsychological Development and Executive Functioning of Children Born to HIV- Infected Mothers
Brief Title: Neuropsychological Development and Executive Functioning of Children Born to HIV- Infected Mothers ( NEUROPSY-HEU )
Acronym: NEUROPSY-HEU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC19_0052
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections; Exposure During Pregnancy; Neurophysiologic Abnormality; Executive Dysfunction
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV exposed children during pregnancy (Experimental): children born from HIV-infected mother, exposed to antiretroviral drugs during pregnancy and in the neonatal period; aged 3 years-old +/- 3 months on the date of inclusion. Parents mastering french language
  Interventions: Diagnostic Test: BRIEF SCORE AT INCLUSION
- control children (Other): children, aged 3 years +/- 3 months on the date of inclusion, from the same socio-economic and cultural environment, not infected or affected by HIV. Parents mastering French language.
  Interventions: Diagnostic Test: BRIEF SCORE AT INCLUSION

INTERVENTIONS:
Diagnostic Test: BRIEF SCORE AT INCLUSION — BRIEF SCALE evaluation

SUMMARY:
Main objective: to evaluate the executive functioning of the HIV exposed uninfected children (HEU) versus children from the same socio-economic and cultural environment, not infected or affected by HIV.

Secondary objective (s): to evaluate Intellectual Quotient, Child development, Behavior, Language and investigate link between executive functioning disorders, exposure to ARVs, HIV and family environment.

DETAILED DESCRIPTION:
The objective of the study is the exploration of executive functions (EF) and screening for neurodevelopment and learning disorders in children born to HIV-infected mothers, exposed to the virus and to antiretrovirals (ARVs).

The evaluation of the executive functioning will be done by the score obtained at the preschool BRIEF for patients and control group issued from questionnaires filled by the mothers of the cases and the mothers of the controls, with matching on age, sex, level of parental education and socio-economic and cultural environment.

Within the group of exposed children, factors associated with executive dysfunction including HIV infection, antiretroviral exposure, maternal socio-demographic data, sociocultural and environmental level will be investigated.

Evolution of the scores between J0, M12 and M24 will be compared within the group of exposed children.

Compared with a control group, the child's intelligence quotient, overall development, behavior and language will be compared at each follow-up time (D0, M12 and M24).

ELIGIBILITY:
Inclusion Criteria:

* experimental:

  * HIV-positive children born to mothers living with HIV antiretrovirals during pregnancy and in the neonatal period, aged 3 years +/- 3 months on the date of inclusion.
  * Parents mastering the French.
* control:

  * children, aged 3 years +/- 3 months on the date of inclusion, from the same socio-economic and cultural environment, no infected or affected by HIV.
  * Parents mastering French.

Exclusion Criteria:

* great prematurity (28-32 weeks)
* genetic anomaly

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
evaluate the executive function of children HEU | inclusion
  Behaviour rating inventary of executive function (BRIEF) preschool version score

SECONDARY OUTCOMES:
Intellectual quotient | at INCLUSION, 12 months after inclusion, 24 months after inclusion
  Wechsler tests score
functional development | at INCLUSION, 12 months after inclusion, 24 months after inclusion
  age and stage questionnaires score
behaviour | at INCLUSION, 12 months after inclusion, 24 months after inclusion
  Strengths and Difficulties Questionnaire score
language | 12 months after inclusion,
  language dysfunction scale score

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Chu Angers, Angers
  - Chd Vendee, La Roche-sur-Yon
  - Chu de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: Undecided